CLINICAL TRIAL: NCT02900053
Title: Post-traumatic Stress Disorder Treatment Using Transcranial Direct Current Stimulation (tDCS) Enhancement of Trauma-focused Therapy : a Two-arm Randomized Controlled Multicentric Study - T-TREAt
Brief Title: Post-traumatic Stress Disorder Treatment Using Transcranial Direct Current Stimulation (tDCS) Enhancement of Trauma-focused Therapy : a Two-arm Randomized Controlled Multicentric Study.
Acronym: T-TREAt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PHRI15-JBC/T-TREAt
Record Dates: First submitted 2016-09-09; First posted 2016-09-14 (Estimated); Last update posted 2025-12-26 (Actual); Status verified 2022-05

CONDITIONS: Post-traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator): Cerebral modulation using tDCS (transcranial Direct-Current Stimulation) associated with repetitive traumatic exposure using a personal traumatic script
  Interventions: Device: tDCS
- Arm 2 (Placebo Comparator): Placebo cerebral modulation using sham-tDCS associated with repetitive traumatic exposure using a personal traumatic script
  Interventions: Device: Placebo tDCS

INTERVENTIONS:
Device: tDCS — tDCS for transcranial Direct-Current Stimulation
  Arms: Arm 1
Device: Placebo tDCS — Placebo tDCS for transcranial Direct-Current Stimulation
  Arms: Arm 2

SUMMARY:
Post-Traumatic Stress Disorder (PTSD) is an anxiety disorder that can develop after exposure to a terrifying event or ordeal in which there was the potential for or actual occurrence of grave physical harm. Traumatic events that may trigger PTSD include violent personal assaults, natural or human-caused disasters, accidents, and military combat. People with PTSD have persistent frightening thoughts and memories of their ordeal, may experience sleep problems, feel detached or numb, or be easily startled. Its lifetime prevalence is quite high, with 7-8% in various studies and 4% in french studies.

The current PTSD treatment usually involves antidepressants as serotonin-specific reuptake inhibitors (SSRIs) and Cognitive Behavioral Therapies, such as exposure therapy to trauma-linked elements (memories, feelings and thoughts) so the fear associated to the traumatic event can decrease. But the therapeutic response stays partial, even combining these treatments.

To improve the PTSD treatment efficiency, innovative approaches are being explored like new drugs or cerebral stimulation. This project aims to assess the efficacy of a less known but promising therapeutic strategy for PTSD : the use of transcranial Direct-Current Stimulation (tDCS) to enhance the trauma-focused therapy results.

ELIGIBILITY:
Inclusion Criteria:

* Having a chronic PTSD (for more than 3 months and less than 10 years) without modification of SSRI long-term treatment for more than 4 weeks
* Between 18 and 65 years-old
* Effective contraception for women, or inability of procreate because of medical or surgical reasons
* Able to give his written informed consent
* Affiliation to a social security system
* Not participating to another study with psychoactive substance

Exclusion Criteria:

* Partially-sighted or partially deaf person requiring equipment
* Person with brain injury or neurological disease (epileptic, tumoral, vascular, degenerative), diagnoses in personal history or recognized as hereditary
* Addiction to psychoactive substance for the last 6 months
* Any treatment which could interact with tDCS effects on cortical reactivity (citalopram, amphetamine, L-dopa, sulpiride, pergolide, lorazepam, rivastigmine, dextromethorphan or other N-methyl-D-aspartate (NMDA) receptor antagonists, d-cycloserine, carbamazepine, flunarizine, calcium channel blockers)
* Pregnancy and lactation
* Any intracephalic metallic material
* Person who can't conform to tests instructions
* Person suffering from bipolar disorder, chronic or acute delusional disorder
* Any circumstances making the person unable to understand the trial features, purposes or consequences

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Evolution of PTSD symptoms | between initial evaluation at J0 before beginning of treatment and follow-up evaluation at 3 month after the end of treatment
  Evolution of PTSD symptoms defined by difference of PTSD severity score measured by Clinician Administered PTSD Scale ( CAPS-5, structured interview)

SECONDARY OUTCOMES:
Evolution of PTSD severity score | between initial evaluation at J0 before beginning of treatment and follow-up evaluation at 1 month after the end of treatment
  Evolution of PTSD severity score (measured with CAPS-5) between initial evaluation at J0 before beginning of treatment and follow-up evaluation at 1 month after the end of treatment
Evolution of PTSD severity score | between initial evaluation at J0 before beginning of treatment, follow-up evaluation at 1 month, follow-up evaluation at 3 month after the end of treatment
  Evolution of PTSD severity score, measured by an auto-questionnaire (PTSD Checklist or Post-Traumatic CheckList Scale (PCL-5)), between initial evaluation at J0 before beginning of treatment, follow-up evaluation at 1 month, follow-up evaluation at 3 month after the end of treatment
Evolution of severity of different PTSD under-dimensions | between initial evaluation at J0 before beginning of treatment, follow-up evaluation at 1 month, follow-up evaluation at 3 month after the end of treatment
  Evolution of severity of different PTSD under-dimensions (intrusive symptoms, evasion symptoms, mood and cognitive symptoms, reactivity and activation symptoms) as measured by CAPS-5 (structured interview) and PCL-5 (auto-questionnaire) between initial evaluation at J0 before beginning of treatment, follow-up evaluation at 1 month, follow-up evaluation at 3 month after the end of treatment
Evolution of comorbid depressive symptoms | between initial evaluation at J0 before beginning of treatment, follow-up evaluation at 1 month, follow-up evaluation at 3 month after the end of treatment
  Evolution of comorbid depressive symptoms measured by Beck depression inventory (BDI), abridged version ; auto-questionnaire) between initial evaluation at J0 before beginning of treatment, follow-up evaluation at 1 month, follow-up evaluation at 3 month after the end of treatment
Evolution of comorbid anxious symptoms | between initial evaluation at J0 before beginning of treatment, follow-up evaluation at 1 month, follow-up evaluation at 3 month after the end of treatment
  Evolution of comorbid anxious symptoms measured by avec la State-Trait Anxiety Inventory (STAI-A ; auto-questionnaire) between initial evaluation at J0 before beginning of treatment, follow-up evaluation at 1 month, follow-up evaluation at 3 month after the end of treatment
Evolution of quality of life symptoms | between initial evaluation at J0 before beginning of treatment, follow-up evaluation at 1 month, follow-up evaluation at 3 month after the end of treatment
  Evolution of quality of life symptoms as measured by World Health Organization Quality Of Life abridged version (WHOQOL-BREF ; auto-questionnaire) between initial evaluation at J0 before beginning of treatment, follow-up evaluation at 1 month, follow-up evaluation at 3 month after the end of treatment
Evolution of quality of life symptoms | between initial evaluation at J0 before beginning of treatment, follow-up evaluation at 1 month, follow-up evaluation at 3 month after the end of treatment
  Evolution of quality of life symptoms as measured by Global Functioning Evaluation scale (EGF) between initial evaluation at J0 before beginning of treatment, follow-up evaluation at 1 month, follow-up evaluation at 3 month after the end of treatment
Evolution of cognitive functioning | between initial evaluation at J0 before beginning of treatment, follow-up evaluation at 1 month, follow-up evaluation at 3 month after the end of treatment
  Evolution of cognitive functioning as measured by Stroop test with emotional variant and n-back test between initial evaluation at J0 before beginning of treatment, follow-up evaluation at 1 month, follow-up evaluation at 3 month after the end of treatment
Evolution of physiological response | between evaluation at rest before the first session, during the first and the last session of tDCS, and 3 months after the last session of treatment
  Evolution of physiological response as measured by cutaneous conductance and cardiac and respiratory frequencies between evaluation at rest before the first session, during the first and the last session of tDCS, and 3 months after the last session of treatment
Evolution of clinical tolerance | After each session
  Evolution of clinical tolerance to this therapeutic procedure by Brunoni questionnaire (nausea, headache, rash, skin redness, tingling, dizziness)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Baptiste Courtine, MD, Principal Investigator — CHRU TOURS
Locations (5):
- France (5):
  - CHU Angers, Angers
  - CHU Nantes, Nantes
  - CHU Poitiers, Poitiers
  - CHU Rennes, Rennes
  - CHU Tours, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Eyraud N, Poupin P, Legrand M, Caille A, Sauvaget A, Bulteau S, Gohier B, Harika-Germaneau G, Drapier D, Jaafari N, Bodic O, Brizard B, Gissot V, Belzung C, Courtine JB, El-Hage W. Combining trauma script exposure with tDCS to alleviate symptoms of posttraumatic stress disorder: A two-arm randomized sham-controlled multicenter trial. Brain Stimul. 2024 May-Jun;17(3):591-593. doi: 10.1016/j.brs.2024.04.018. Epub 2024 May 3. No abstract available. PMID 38704084